CLINICAL TRIAL: NCT00540605
Title: Phase I Study of the Maternal Single-Dose Pharmacokinetics and Placental Transfer of Tenofovir 1% Vaginal Gel Among Healthy Term Gravidas
Brief Title: Blood Levels of Tenofovir Gel in HIV Uninfected Pregnant Women Planning Cesarean Delivery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Microbicide Trials Network (Network); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MTN-002; 10600 (Registry Identifier: DAIDS ES); 1-U01-AI068633-0; 1U01AI068633 (NIH); NCT00572273 (obsolete NCT alias)
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2012-05

CONDITIONS: HIV Infections
Keywords: Microbicide; Pregnancy; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): 4g tenofovir 1% gel applied vaginally 2 hours prior to expected time of cesarean delivery
  Interventions: Drug: Tenofovir 1% vaginal gel

INTERVENTIONS:
Drug: Tenofovir 1% vaginal gel — topical gel containing 1% tenofovir

SUMMARY:
A new approach to HIV prevention currently being studied includes the use of topical microbicides, substances that kill microbes. The purpose of this study is to determine the levels of tenofovir, a microbicide in gel form, in HIV uninfected pregnant women who are expecting to deliver by cesarean.

DETAILED DESCRIPTION:
There is an urgent need for HIV prevention methods that women can initiate and control themselves. Topical microbicides represent one such method. Tenofovir 1% vaginal gel was chosen as a high priority microbicide candidate due to its activity in target cells for HIV infection of the vagina and cervix and the low frequency of local and systemic toxicity observed in a prior HIV Prevention Trials Network (HPTN) trial utilizing tenofovir 1% gel. The purpose of this study is to assess term pregnancy single-dose pharmacokinetics (PK) of tenofovir 1% gel in HIV uninfected pregnant women.

The expected duration of participation for individually enrolled participants will depend on how early they enroll prior to the date of cesarean section, but may range from approximately 3 to 6 weeks. An initial screening/enrollment visit will occur approximately 1 to 4 weeks prior to the participant's scheduled cesarean section, but no more than 4 weeks before the delivery date. A targeted physical exam, medical and medication history assessment, blood and urine collection, and a pelvic exam will occur at screening/enrollment. Tenofovir gel will be administered vaginally approximately 2 hours before the expected time of cesarean section. On the day of gel administration and cesarean delivery, a targeted physical exam, medical and medication history assessment, a pelvic exam, maternal blood tenofovir level measurement, and collection of placental and endometrial tissues, cord blood, and amniotic fluid will occur.

After gel administration, PK measures will be taken at Hours 1, 2, 4, 6, 8, and 12; maternal blood tenofovir level measurement and a review of adverse events will also occur at these times. A 24-hour evaluation will occur between Hours 22 and 26. At this evaluation, a targeted physical exam, a review of adverse events, and tenofovir level measurement will occur. Each participant will be contacted between Days 10 and 18 to collect data on any adverse events they experience. In addition, an unscheduled visit may be necessary if an unresolved adverse event occurs on or after the 24-hour evaluation. If an unscheduled visit is required, the participant will undergo a targeted physical exam, medical and medication history assessment, blood and urine collection, a pelvic exam, and tenofovir level measurement.

ELIGIBILITY:
Inclusion Criteria:

* General good health
* HIV uninfected
* Hepatitis B surface antigen negative at screening and enrollment
* Viable, single pregnancy delivered by cesarean section planned between 37 0/7 to 41 6/7 weeks of pregnancy
* Normal Pap smear in the 12 months prior to study entry
* Willing to abstain from vaginal, anal, and receptive oral sex for at least 2 weeks after gel administration
* Willing to abstain from intravaginal products and practices (including douching) during study participation

Exclusion Criteria:

* Maternal or fetal condition that requires urgent cesarean section
* Documented rupture of the amniotic membranes
* Known disease in the mother that has a predictable negative effect on placental function
* Known placental/fetal abnormalities that could affect placental transfer. More information on this criterion can be found in the protocol.
* Previously demonstrated hypersensitivity to any components of tenofovir 1% gel
* Certain abnormal laboratory values
* Use of vaginal medications within 48 hours of study entry
* Untreated sexually transmitted infection (STI) or exposure to partner's STI, including chlamydia, gonorrhea, trichomoniasis, and nongonococcal urethritis
* Symptomatic vaginitis, including bacterial vaginosis and vulvovaginal candidiasis. Participants with asymptomatic signs of bacterial vaginosis and/or yeast not excluded.
* Participation in any other investigational drug or device trial within 30 days of study entry
* Any social or medical condition that, in the opinion of the investigator, would interfere with the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Maternal third trimester pharmacokinetic (PK) measures (AUC and Cmax) | Throughout study
Endometrial tenofovir levels | At Hours 1, 2, 4, 6, 8, 12, and 24 after drug administration
Placental transfer (cord blood tenofovir levels, placental tissue tenofovir levels, and amniotic fluid tenofovir levels) | At Hours 1, 2, 4, 6, 8, 12, and 24 after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Richard Beigi, MD, MSc, FACOG, Study Chair — Magee-Women's Hospital of UPMC, Department of Obstetrics/Gynecology; Sharon Hillier, PhD, Principal Investigator — Microbicides Trial Network
Locations (1):
- Pitt CRS, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Carballo-Dieguez A, Balan IC, Morrow K, Rosen R, Mantell JE, Gai F, Hoffman S, Maslankowski L, El-Sadr W, Mayer K. Acceptability of tenofovir gel as a vaginal microbicide by US male participants in a Phase I clinical trial (HPTN 050). AIDS Care. 2007 Sep;19(8):1026-31. doi: 10.1080/09540120701294237. PMID 17852000
- [Background] Mayer KH, Maslankowski LA, Gai F, El-Sadr WM, Justman J, Kwiecien A, Masse B, Eshleman SH, Hendrix C, Morrow K, Rooney JF, Soto-Torres L; HPTN 050 Protocol Team. Safety and tolerability of tenofovir vaginal gel in abstinent and sexually active HIV-infected and uninfected women. AIDS. 2006 Feb 28;20(4):543-51. doi: 10.1097/01.aids.0000210608.70762.c3. PMID 16470118
- [Derived] Beigi R, Noguchi L, Parsons T, Macio I, Kunjara Na Ayudhya RP, Chen J, Hendrix CW, Masse B, Valentine M, Piper J, Watts DH. Pharmacokinetics and placental transfer of single-dose tenofovir 1% vaginal gel in term pregnancy. J Infect Dis. 2011 Nov 15;204(10):1527-31. doi: 10.1093/infdis/jir562. Epub 2011 Sep 19. PMID 21930612